CLINICAL TRIAL: NCT00163462
Title: Comparison of Ciclesonide (80 mcg or 160 mcg Once Daily in the Evening) and Fluticasone Propionate (100 mcg Twice Daily in the Morning and Evening) in Pediatric Asthma Patients
Brief Title: Efficacy of Ciclesonide Inhaled Once Daily Versus Fluticasone Propionate Inhaled Twice Daily in Children With Asthma (6 to 11 y) (BY9010/M1-206)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BY9010/M1-206
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-10

CONDITIONS: Asthma
Keywords: Asthma; Ciclesonide; Child; Fluticasone propionate; Pediatric
MeSH Terms: conditions — Asthma | interventions — ciclesonide

INTERVENTIONS:
Drug: Ciclesonide

SUMMARY:
The aim of the study is to compare the efficacy of ciclesonide versus fluticasone propionate on lung function, symptoms, and use of rescue medication in children with persistent asthma. Ciclesonide will be inhaled once daily, using one of the two dose levels; fluticasone propionate will be inhaled at one dose level twice daily. The study duration consists of a baseline period (2 to 4 weeks) and a treatment period (12 weeks). The study will provide further data on safety and tolerability of ciclesonide.

ELIGIBILITY:
Main Inclusion Criteria:

* History of persistent bronchial asthma for at least 6 months
* FEV1 50-90% of predicted

Main Exclusion Criteria:

* Concomitant severe diseases or diseases which are contraindications for the use of inhaled steroids
* COPD (chronic bronchitis or emphysema) and/or other relevant lung diseases causing alternating impairment in lung function
* Respiratory tract infection or asthma exacerbation within the last 30 days prior to entry into the study
* History of life-threatening asthma
* Premature birth
* Current smoking
* Smoking history with either equal or more than 10 pack-years
* Pregnancy
* Intention to become pregnant during the course of the study
* Breast feeding
* Lack of safe contraception

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 750
Dates: Start 2004-10; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
FEV1 absolute values
PD20FEV1 from methacholine challenge.

SECONDARY OUTCOMES:
FEV1 as % of predicted
PEF from spirometry
morning and evening PEF from diary
asthma symptom score from diary
salbutamol MDI use from diary
diurnal PEF fluctuation from diary
dropout rate due to asthma exacerbations and time to the first asthma exacerbation
percentage of asthma symptom-free days, rescue medication-free days, nocturnal awakening free days and days on which patients perceived asthma control
onset of effect assessed by morning PEF, asthma total symptom score and use of rescue medication
interview administered PAQLQ(S), self-administered PACQLQ
physical examination and vital signs
laboratory investigation
AEs
HPA-axis function assessed by free cortisol concentration in 24 hour-urine samples.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (48):
- Brazil (10):
  - Altana Pharma/Nycomed, Campinas - SP
  - Altana Pharma/Nycomed, Curitiba-PR
  - Altana Pharma/Nycomed, Florianópolis-SC
  - Altana Pharma/Nycomed, Porto Alegre-RS
  - Altana Pharma/Nycomed, Rio de Janeiro-RJ
  - Altana Pharma/Nycomed, Salvador - Bahia
  - Altana Pharma/Nycomed, Santo André-SP
  - Altana Pharma/Nycomed, Sao Paulo - SP
  - Altana Pharma/Nycomed, Sao Paulo-SP
  - Altana Pharma/Nycomed, São Paulo-SP
- Germany (7):
  - Altana Pharma/Nycomed, Frankfurt
  - Altana Pharma/Nycomed, Gaißach Bei Bad Tölz
  - Altana Pharma/Nycomed, Geesthacht
  - Altana Pharma/Nycomed, Mainz
  - Altana Pharma/Nycomed, München
  - Altana Pharma/Nycomed, Wesel
  - Altana Pharma/Nycomed, Wiefelstede
- Hungary (7):
  - Altana Pharma/Nycomed, Budapest
  - Altana Pharma/Nycomed, Debrecen
  - Altana Pharma/Nycomed, Jászberény
  - Altana Pharma/Nycomed, Miskolc
  - Altana Pharma/Nycomed, Mosdós
  - Altana Pharma/Nycomed, Pécs
  - Altana Pharma/Nycomed, Törökbálint
- Poland (7):
  - Altana Pharma/Nycomed, Inowrocław
  - Altana Pharma/Nycomed, Lodz
  - Altana Pharma/Nycomed, Lublin
  - Altana Pharma/Nycomed, Poznan
  - Altana Pharma/Nycomed, Rzeszów
  - Altana Pharma/Nycomed, Warsaw
  - Altana Pharma/Nycomed, Zawadzkie
- Portugal (10):
  - Altana Pharma/Nycomed, Amadora
  - Altana Pharma/Nycomed, Faro
  - Altana Pharma/Nycomed, Guimarães
  - Altana Pharma/Nycomed, Lisbon
  - Altana Pharma/Nycomed, Matosinhos Municipality
  - Altana Pharma/Nycomed, Oliveira de Azeméis
  - Altana Pharma/Nycomed, Porto
  - Altana Pharma/Nycomed, Setúbal
  - Altana Pharma/Nycomed, Viana do Castelo
  - Altana Pharma/Nycomed, Vila Nova de Gaia
- South Africa (7):
  - Altana Pharma/Nycomed, Bellville - Cape Town -
  - Altana Pharma/Nycomed, Cape Town
  - Altana Pharma/Nycomed, Morningside, Sandton
  - Altana Pharma/Nycomed, Mowbray, Cape Town
  - Altana Pharma/Nycomed, Panorama / RSA-Cape Town
  - Altana Pharma/Nycomed, Westville
  - Altana Pharma/Nycomed, Wynberg

REFERENCES:
- See also: BY9010-MI-206-RDS-2006-09-01.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4526&filename=BY9010-MI-206-RDS-2006-09-01.pdf